CLINICAL TRIAL: NCT02179827
Title: The Evaluation of Minimally Invasive Hemodynamic Monitors for the Assessment of Volume Responsiveness to Various Standard Replacement Fluids During Acute Normovolemic Hemodilution
Brief Title: Performance of Non-Invasive Monitors During ANH
Status: Withdrawn | Type: Observational
Why Stopped: Study never commenced, and is now closed.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 362559
Record Dates: First submitted 2014-03-11; First posted 2014-07-02 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Baseline; Hemodilution

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to assess the responsiveness of the standard minimally invasive hemodynamic monitors used in the operating room to known changes in the intravascular volume status that occur during blood removal and volume replacement with three different standard fluids used during ANH.

ELIGIBILITY:
Inclusion Criteria:

* Those surgical procedures where ANH is included in the surgical plan and consent is obtained

Exclusion Criteria:

* Severe or symptomatic COPD, emphysema, renal, hepatic or coronary artery disease as defined by the American College of Cardiology (Cannon et al., 2001).
* Esophageal pathology (diverticulum, hiatal hernia, esophageal cancer, esophageal surgery), which introduces risks associated with the placement of the esophageal Doppler.
* Ascites.
* BMI >35
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective procedures requiring normovolemic hemodilution
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac output | Baseline (Supine) Volume Replaced (S/P ANH)
  Metrics: Cardiac output stroke volume Stroke volume: variation

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Health System, Sacramento, California, United States